CLINICAL TRIAL: NCT02003417
Title: A Multicenter Study to Evaluate Cardiovascular Risk Factors and Receipt of Primary and Preventive Care in Prostate Cancer Patients Who Receive Definitive Radiation Therapy and Androgen Deprivation Therapy.
Brief Title: Cardiovascular Risk and Preventive Care in Prostate Cancer Patients Receiving Radiation and Hormone Therapy
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Radiation Therapy Oncology Group (Network)
Responsible Party: Sponsor
Other Study IDs: LCCC 1218
Record Dates: First submitted 2013-11-18; First posted 2013-12-06 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; External beam radiation treatment; Androgen deprivation therapy; Definitive treatment; Cardiovascular risk factors; Quality of life
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Non-metastatic prostate cancer patients: Histologically-confirmed, non-metastatic prostate cancer patients who received external beam radiation treatment with androgen deprivation therapy (total ADT duration > 3 months) for definitive treatment.

SUMMARY:
This study will evaluate the proportion of prostate cancer patients receiving external beam radiation therapy (EBRT) and androgen deprivation therapy (ADT) with controlled blood sugars (fasting glucose and hemoglobin A1c), blood pressure, and cholesterol profile (total cholesterol, LDL, HDL, triglycerides) at baseline, 3 months, and 12 months after completing radiation treatment. In addition, receipt of guideline-recommended cardiovascular, primary and preventive care as well as patient-reported quality of life and satisfaction with care among these patients will be evaluated at baseline and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed, non-metastatic prostate cancer
* Patients who will receive external beam radiation treatment with androgen deprivation therapy (total ADT duration > 3 months) for curative treatment, either in the definitive or post-prostatectomy setting
* Patients who have a primary care provider
* Informed consent obtained and signed
* Ability to read and write English
* Age >= 18
* No mental incompetence which would preclude completion of questionnaires

Exclusion Criteria:

* Prior cancer, pelvic radiation treatment or chemotherapy
* Patients who do not have a primary care provider
* Prior ADT
* Mental incompetence which would preclude completion of questionnaires
* Unable to read and write English

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically-confirmed, non-metastatic prostate cancer patients who visit radiation oncology clinics at participating institutions: The University of North Carolina at Chapel Hill Cancer Hospital, Rex Cancer Center at the Raleigh and Wakefield locations, Marion J. Shepard Cancer Center, Coastal Carolina Radiation Oncology, The University of Virginia, High Point Regional UNC Health Care, and MedStar Georgetown University. Patients with planned radiation treatment and androgen deprivation therapy with curative intent (in definitive or post-prostatectomy settings) are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2012-06; Primary Completion 2016-07 (Actual); Study Completion 2018-05-04 (Actual)

PRIMARY OUTCOMES:
Proportion of prostate cancer patients with controlled blood sugars, blood pressure, and cholesterol profile. | Baseline
  Blood sugars include fasting glucose and hemoglobin A1c; blood pressure includes systolic and diastolic; and cholesterol profile includes total cholesterol, LDL, HDL, and triglycerides. Baseline is prior to receiving androgen deprivation therapy and prior to radiation.

SECONDARY OUTCOMES:
Proportion of prostate cancer patients with controlled blood sugars, blood pressure, and cholesterol profile. | 3 months post radiation treatment completion
  Blood sugars include fasting glucose and hemoglobin A1c; blood pressure includes systolic and diastolic; and cholesterol profile includes total cholesterol, LDL, HDL, and triglycerides.
Proportion of prostate cancer patients with controlled blood sugars, blood pressure, and cholesterol profile. | 12 months post radiation treatment completion
  Blood sugars include fasting glucose and hemoglobin A1c; blood pressure includes systolic and diastolic; and cholesterol profile includes total cholesterol, LDL, HDL, and triglycerides.
Proportion of prostate cancer patients with guideline-recommended cardiovascular preventive care (glucose testing, cholesterol testing, and blood pressure measurement). | Baseline
  This will be done by patient self-report and by medical record review (radiation oncologist will obtain medical records from patient's primary care physician).
Proportion of prostate cancer patients with guideline-recommended cardiovascular preventive care (glucose testing, cholesterol testing, and blood pressure measurement). | 12 months post radiation treatment completion
  This will be done by patient self-report and by medical record review (radiation oncologist will obtain medical records from patient's primary care physician).
Proportion of prostate cancer patients who receive other (non-cardiovascular) guideline-recommended primary and preventive care (flu vaccination, colorectal cancer screening, and healthy lifestyle counseling). | Baseline
  This will be done by patient self-report and by medical record review (radiation oncologist will obtain medical records from patient's primary care physician).
Proportion of prostate cancer patients who receive other (non-cardiovascular) guideline-recommended primary and preventive care (flu vaccination, colorectal cancer screening, and healthy lifestyle counseling). | 12 months post radiation treatment completion
  This will be done by patient self-report and by medical record review (radiation oncologist will obtain medical records from patient's primary care physician).
Patient-reported quality of life. | Baseline
Patient-reported quality of life. | 12 months post radiation treatment completion
Patient-reported coordination of care. | Baseline
Patient-reported coordination of care. | 12 months post radiation treatment completion
Patient-reported satisfaction with care. | Baseline
Patient-reported satisfaction with care. | 12 months post radiation treatment completion

CONTACTS AND LOCATIONS:
Overall Officials: Ronald C Chen, MD, MPH, Principal Investigator — University of North Carolina at Chapel Hill - Department of Radiation Oncology
Locations (8):
- United States (8):
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - University of North Carolina at Chapel Hill Cancer Hospital, Chapel Hill, North Carolina
  - High Point Regional UNC Health Care, High Point, North Carolina
  - Rex Healthcare, Inc, Raleigh, North Carolina
  - Rex Healthcare of Wakefield, Raleigh, North Carolina
  - Marion L. Shepard Cancer Center, Washington, North Carolina
  - Coastal Carolina Radiation Oncology, Wilmington, North Carolina
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center — http://unclineberger.org/
- See also: National Cancer Institute — http://www.cancer.gov/